CLINICAL TRIAL: NCT05195203
Title: A Phase I Randomized, Double-blinded, Placebo-controlled Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetic of HS-10353 in Chinese Adult Subjects
Brief Title: A Study of HS-10353 in Chinese Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10353-101
Record Dates: First submitted 2021-08-12; First posted 2022-01-18 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Major Depressive Disorder
Keywords: Phase I; major depressive disorder; healthy subject; SAD; MAD
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10353 (Experimental): Capsules；Single dose: only one administration; Multiple doses: continuous administration for 7 days
  Interventions: Drug: HS-10353
- Placebo (Placebo Comparator): Capsules；Single dose: only one administration; Multiple doses: continuous administration for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HS-10353 — Single or multiple dose(s) of HS-10353
  Other Names: HS-10353 capsules
  Arms: HS-10353
Drug: Placebo — Single or multiple dose(s) of placebo
  Other Names: HS-10353 placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of single and multiple oral administered doses of HS-10353 separately in Chinese healthy and major depressive disorder subjects.

DETAILED DESCRIPTION:
This is a phase I, randomized, double-blinded, placebo-controlled, both single ascending doses (SAD) study and multiple ascending dose (MAD) clinical trial to assess the safety, tolerability, and pharmacokinetics of HS-10353 tablet(s) separately in Chinese healthy and major depressive disorder (MDD) subjects.

Approximately six sequential dose cohorts will be evaluated in SAD study. Sentinel dosing will be employed for the first SAD cohort to protect the subjects' safety. Escalation to the next dose cohort will be undertaken only after safety and PK data are reviewed by the Safety Review Committee (SRC) and agreement reach that it is safe to increase the dose. Each SAD cohort is dosed at approximately weekly intervals to allow adequate time for collection and review of safety and PK data.

Approximately three sequential dose cohorts will be evaluated in MAD study. The total daily dose for each MAD cohort will be based on information obtained from the SAD study. Each subject will receive only one dose regimen in this study.

Safety data up to Day14 (±1) in SAD and up to Day20 (±1) in MAD will be reviewed prior to the next dose level. The number of Cohorts in SAD and MAD would be adjusted based on the assessment of SRC.

ELIGIBILITY:
SAD Inclusion Criteria

1. Healthy male or female subjects between 18 and 45 years old;
2. Body weight more than 50.0kg (male) or 45.0kg (female), body mass index (BMI) within the range of 19.0~26.0kg/m2;
3. Volunteers agree to refrain from smoking, drinking alcohol. Avoid xanthine or caffeine (including chocolate, tea, coffee, cola, etc.) and avoid strenuous exercise;
4. The male volunteers agreed to refrain from donating sperm from the start of the drug until six months after they stopped the study;
5. The female volunteers agreed to avoid ovum donation from the start of the drug until six months after they stopped the study;
6. Pregnancy test results of female volunteers must be negative within 3 days of administration.

SAD Exclusion Criteria

1. Pregnant and breastfeeding female.
2. Volunteers with a history of cardiovascular, respiratory, liver, kidney, digestive tract, mental, neurological, hematological, metabolic and other systemic diseases, who are not suitable to participate in this study as assessed by the investigator.
3. The results of vital signs, physical examination, laboratory examination and 12-lead ECG during screening were abnormal with clinical significance.
4. Hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), human immunodeficiency virus antibody (HIVAb) or syphilis antibody is positive
5. Volunteers had a history of drug dependence or abuse.
6. A heavy smoker or smokers who smoked 5 or more cigarettes per day for 3 months prior to screening or tested positive for nicotine during screening.
7. A history of alcohol abuse or a single consumption of more than 14 units of alcohol (1 unit = 285 mL of beer, 25 mL of spirits, 150 mL of wine) in the nearly two weeks prior to screening or a positive breath test for alcohol at screening.
8. Participate in clinical trials of any drug or medical device within 3 months prior to screening.
9. Any medication taken within 2 weeks of administration, including prescription, over-the-counter, and herbal medicines.
10. Diet or dietary treatment or significant change in dietary habits within 30 days prior to administration for whatever reason.
11. Volunteers who have difficulty swallowing solid tablets or capsule.
12. Volunteers with difficulty in blood collection, unable to tolerate multiple venous blood collection and any blood collection contraindications.

MAD Inclusion Criteria

1. Subject has signed an ICF prior to any study-specific procedures being performed.
2. Subject is an ambulatory male or female between 18 and 65 years of age, inclusive.
3. Subject has a diagnosis of MDD that has been present for at least a 4-week period as diagnosed by DSM-5.
4. Subject has a HAM-D17 total score of ≥22 at screening and Day 1 (prior to dosing).
5. Subject is willing to discontinue other antidepressant or anti-anxiety medications （such as benzodiazepines） or antipsychotics during screening and treatment.

MAD Exclusion criteria:

1. Subject has a history of suicide attempt.
2. Subject has a recent history or active clinically significant manifestations of metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, musculoskeletal, dermatological, urogenital, neurological, or eyes, ears, nose, and throat disorders, or any other acute or chronic condition that, in the Investigator's opinion, would limit the subject's ability to complete or participate in this clinical study.
3. Subject has a history of treatment-resistant depression, defined as persistent depressive symptoms despite treatment with adequate doses of antidepressants from two different classes for an adequate amount of time (ie, at least 4 weeks of treatment).
4. Subject has detectable hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV), or human immunodeficiency virus (HIV) antibody at screening.
5. Subject has active psychosis per Investigator assessment.
6. Subject has a medical history of seizures.
7. Subject has a medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder.
8. Subject has had exposure to another investigational medication or device within 30 days prior to screening.
9. Subject has had administration of psychotropics that have been initiated within 14 days prior to screening and/or are not being taken at a stable dose.
10. Use of any known strong inhibitors and/or inducers of cytochrome P450 (CYP)3A4 within the 14 days or five half-lives (whichever is longer) or consumed grapefruit juice, grapefruit, Seville oranges, or products containing these within 30 days prior to receiving the first dose of study drug.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-03-11 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Endpoints of the trial：AE，SAE | Baseline to end of follow-up (a maximum of 20 days)
  The incidence, severity, and association of AE, SAE and AE leading to withdrawal from the trial

SECONDARY OUTCOMES:
SAD pharmacokinetic endpoints：Cmax | Day1-Day6
  The maximum plasma concentration (Cmax)
SAD pharmacokinetic endpoints：Tmax | Day1-Day6
  Time to Cmax (Tmax)
SAD pharmacokinetic endpoints：AUC0-t | Day1-Day6
  The area under the plasma concentration-time curve from time zero to the time of the last measurable concentration (AUC0-t)
SAD pharmacokinetic endpoints：AUC0-∞ | Day1-Day6
  The area under the plasma concentration-time curve from time zero to infinite time (AUC0-∞)
SAD pharmacokinetic endpoints：λz | Day1-Day6
  Terminal rate constant (λz)
SAD pharmacokinetic endpoints：t½ | Day1-Day6
  Half-life (t½)
SAD pharmacokinetic endpoints：CL/F | Day1-Day6
  Apparent clearance following oral administration (CL/F)
SAD pharmacokinetic endpoints：Vz/F | Day1-Day6
  Apparent volume of distribution following oral administration (Vz/F)
SAD pharmacokinetic endpoints：MRT | Day1-Day6
  Mean residence time (MRT)
MAD pharmacokinetic endpoints：Css,max | Day1-Day12
  The maximum steady state drug concentration in plasma during dosing interval (Css,max)
MAD pharmacokinetic endpoints：Css,av | Day1-Day12
  Average steady state drug concentration in plasma during dosing interval (Css,av)
MAD pharmacokinetic endpoints：Tss,max | Day1-Day12
  Time to Css, max (Tss,max)
MAD pharmacokinetic endpoints：AUCss, 0-t | Day1-Day12
  The area under the plasma concentration-time curve from time zero to the time of the last measurable concentration over the dosing interval at steady state (AUCss, 0-t)
MAD pharmacokinetic endpoints：DF | Day1-Day12
  Coefficient of fluctuation（DF）
MAD pharmacokinetic endpoints：Rac | Day1-Day12
  Accumulation ratio (Rac)
MAD pharmacokinetic endpoints：Css,min | Day1-Day12
  The minimum steady state drug concentration in plasma during dosing interval (Css,min)

OTHER OUTCOMES:
MAD pharmacodynamics endpoints：Ham-D17 response rate | Day1-Day12
  Ham-D17 response rate (score decreased ≥50% from baseline) and (score ≤7)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Background] Whiteford HA, Degenhardt L, Rehm J, Baxter AJ, Ferrari AJ, Erskine HE, Charlson FJ, Norman RE, Flaxman AD, Johns N, Burstein R, Murray CJ, Vos T. Global burden of disease attributable to mental and substance use disorders: findings from the Global Burden of Disease Study 2010. Lancet. 2013 Nov 9;382(9904):1575-86. doi: 10.1016/S0140-6736(13)61611-6. Epub 2013 Aug 29. PMID 23993280
- [Background] McIntyre RS, Suppes T, Tandon R, Ostacher M. Florida Best Practice Psychotherapeutic Medication Guidelines for Adults With Major Depressive Disorder. J Clin Psychiatry. 2017 Jun;78(6):703-713. doi: 10.4088/JCP.16cs10885. PMID 28682531
- [Background] Papakostas GI, Fava M. Does the probability of receiving placebo influence clinical trial outcome? A meta-regression of double-blind, randomized clinical trials in MDD. Eur Neuropsychopharmacol. 2009 Jan;19(1):34-40. doi: 10.1016/j.euroneuro.2008.08.009. Epub 2008 Sep 26. PMID 18823760
- [Background] Luscher B, Shen Q, Sahir N. The GABAergic deficit hypothesis of major depressive disorder. Mol Psychiatry. 2011 Apr;16(4):383-406. doi: 10.1038/mp.2010.120. Epub 2010 Nov 16. PMID 21079608
- [Background] Mann JJ, Oquendo MA, Watson KT, Boldrini M, Malone KM, Ellis SP, Sullivan G, Cooper TB, Xie S, Currier D. Anxiety in major depression and cerebrospinal fluid free gamma-aminobutyric acid. Depress Anxiety. 2014 Oct;31(10):814-21. doi: 10.1002/da.22278. Epub 2014 May 27. PMID 24865448
- [Background] Schur RR, Draisma LW, Wijnen JP, Boks MP, Koevoets MG, Joels M, Klomp DW, Kahn RS, Vinkers CH. Brain GABA levels across psychiatric disorders: A systematic literature review and meta-analysis of (1) H-MRS studies. Hum Brain Mapp. 2016 Sep;37(9):3337-52. doi: 10.1002/hbm.23244. Epub 2016 May 4. PMID 27145016
- [Background] Zorumski CF, Paul SM, Izumi Y, Covey DF, Mennerick S. Neurosteroids, stress and depression: potential therapeutic opportunities. Neurosci Biobehav Rev. 2013 Jan;37(1):109-22. doi: 10.1016/j.neubiorev.2012.10.005. Epub 2012 Oct 17. PMID 23085210
- [Background] Uzunova V, Sheline Y, Davis JM, Rasmusson A, Uzunov DP, Costa E, Guidotti A. Increase in the cerebrospinal fluid content of neurosteroids in patients with unipolar major depression who are receiving fluoxetine or fluvoxamine. Proc Natl Acad Sci U S A. 1998 Mar 17;95(6):3239-44. doi: 10.1073/pnas.95.6.3239. PMID 9501247
- [Background] Fellmeth G, Fazel M, Plugge E. Migration and perinatal mental health in women from low- and middle-income countries: a systematic review and meta-analysis. BJOG. 2017 Apr;124(5):742-752. doi: 10.1111/1471-0528.14184. Epub 2016 Jun 20. PMID 27320110
- [Background] Osborne LM, Gispen F, Sanyal A, Yenokyan G, Meilman S, Payne JL. Lower allopregnanolone during pregnancy predicts postpartum depression: An exploratory study. Psychoneuroendocrinology. 2017 May;79:116-121. doi: 10.1016/j.psyneuen.2017.02.012. Epub 2017 Feb 16. PMID 28278440